CLINICAL TRIAL: NCT03837171
Title: Stratégie Transfusionnelle érythrocytaire Dans la réanimation du Choc Septique du Patient d'Onco-hématologie : Essai randomisé Multicentrique TRANSPORT [TRANSfusion in Patients With Onco-hematological Malignancies ResusciTated From Septic Shock]
Brief Title: TRANSfusion in Patients With Onco-hematological Malignancies ResusciTated From Septic Shock
Acronym: TRANSPORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K170913J; 2018-A00592-53 (Other: IDRCB)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock; Anemia; Cancer
Keywords: Septic Shock; Anemia; cancer; erythrocyte transfusion
MeSH Terms: conditions — Shock, Septic; Anemia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal strategy (Active Comparator): Maintain a hemoglobin level > 9 g/dL during the first 48 hours of resuscitation of septic shock
  Interventions: Biological: Liberal Red blood cell transfusion
- Restrictive strategy (Experimental): Maintain a hemoglobin level > 7 g/dL during the resuscitation of septic shock
  Interventions: Biological: Restrictive Red blood cell transfusion

INTERVENTIONS:
Biological: Liberal Red blood cell transfusion — Hemoglobin level will be maintained above 9 g/dL (liberal strategy) for the first 48 hours following randomization. After 48 hours, indications of RBC transfusions will be at the discretion of attending physicians in patients with persistent circulatory failure.
  After resolution of acute circulatory failure, a 7 g/dL transfusion threshold will be recommended regardless of the allocation arm. In case of subsequent episodes of septic shock, the transfusion strategy will be at the discretion of attending physicians
  Arms: Liberal strategy
Biological: Restrictive Red blood cell transfusion — Hemoglobin level will be maintained above 7 g/dL (restrictive strategy) during all the stay in ICU
  Arms: Restrictive strategy

SUMMARY:
Septic shock is a frequent complication associated with high mortality in patients with malignancies. The best transfusion strategy (restrictive or liberal) for the resuscitation of septic shock remains a controversial issue, in relation with potentially discrepant goals of tissue oxygenation and transfusion sparing.

In this study, the investigators propose to address the efficacy of two RBC transfusion strategies (liberal or restrictive) in restoring appropriate tissue oxygenation as well as their tolerance.

The investigators designed a prospective randomized multicenter trial aimed at comparing liberal and restrictive RBC transfusion strategies applied during the first 48 hours of resuscitation in cancer patients with septic shock and anemia.

DETAILED DESCRIPTION:
Septic shock is a frequent complication in patients with malignancies and remains affected with a mortality rate higher than 50%.

Red blood cell (RBC) transfusion remains a major issue for critically ill cancer patients who frequently display anemia as a result of malignant bone marrow involvement or imposed by cytotoxic treatments. However, our current practice of RBC transfusion in the intensive care unit (ICU) is drawn from general populations. Several case-control studies suggested that RBC transfusion was associated with higher mortality and increased incidence of ICU-acquired complications in critically ill patients. In 1999, a restrictive strategy of non-leucodepleted RBC transfusion to maintain hemoglobin above 7 g/dL was shown to be as effective as a liberal transfusion strategy aimed to maintain haemoglobin > 10 g/dL in critically ill patients. As of today, the current recommendations for RBC transfusion remain largely based on this study which excluded patients with a history of anemia. Leucodepletion that is now routinely implemented in France might be associated with fewer transfusion-related events. Indeed, some recent studies challenged the restrictive strategy and suggested that a higher transfusion threshold might be beneficial in septic patients for whom oxygen delivery is of paramount importance. Most importantly, a hemodynamic support algorithm for severe sepsis also known as early goal-directed therapy (EGDT) included a hematocrit target of 30%. The majority of EGDT-treated patients received RBC transfusion within the early 72 hours of resuscitation, thereby representing a major difference compared to standard treatment, but the prognostic value of RBC transfusion was not specifically assessed. A recent case-control study also suggested that RBC transfusion was an independent predictor of survival in patients with septic shock.

Cancer patients with septic shock and hemoglobin level < 9 g/dL initiation will be randomized to the interventional arm (liberal transfusion strategy to maintain hemoglobin > 9 g/dL) or to the control arm (restrictive transfusion strategy to maintain hemoglobin > 7 g/dL) in a 1:1 ratio.

Patients from the intervention arm will have their hemoglobin level maintained above 9 g/dL for the whole time under vasopressors, for a maximum of 28 days. After weaning from vasopressor, the transfusion threshold will be lowered to 7 g/dL as recommended by the SSC guidelines. In case of shock relapse requiring reintroduction of vasopressors, the transfusion threshold will be upgraded back to 9 g/dL until next catecholamine weaning.

In the control arm, the transfusion threshold will be 7 g/dL until ICU discharge regardless of catecholamine administration.

The primary objective of the study will be the restoration of tissue oxygenation as assessed by lactate clearance at 12 hours following randomization. The secondary endpoints will be related to restoration of tissue oxygenation at alternative time points (6h, 24h, 36h, 48h) as assessed as above, the 7-day, 28-day, in-ICU and in-hospital mortality rate, changes in organ failures over the first 48 hours and 7 days, duration for organ failure supports, the development of acute ischemic and thrombotic events (myocardial infarction, mesenteric ischemia, ischemic stroke, limb ischemia, deep venous thrombosis) over the first 7 days.

An interim analysis on the primary endpoint has been pre-planned at the end of the follow up of half of patients included.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Evolutive (complete remission < 2 years) malignant solid tumor or chronic or acute hematological malignancy
* Septic shock defined as:
* Presumed or documented infection
* Acute circulatory failure defined as hypotension requirement of vasoactive drugs for more than one hour (norepinephrine or epinephrine ≥ 0.1 µg/kg/min)
* Tissue hypoxia defined by arterial lactate level > 2 mmol/L within 3 hours prior to inclusion
* Hemoglobin level < 9 g/dL
* Informed consent from patients or surrogates

Exclusion Criteria:

* Acute life-threatening bleeding
* Ongoing acute coronary syndrome or any other acute ischemic condition
* End-of-life decisions at the time of ICU admission
* Refusal of transfusions for personal beliefs
* Lack of social security coverage
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation | 12 hours
  Percentage of patients with normal arterial lactate level at 12 hours (<=2 mmol/L) or a relative decrease (or clearance) of arterial lactate level above 30% according to the formula (lactateH0 - lactateH12)/lactate H0*100.
  lactateH0 : arterial lactate level at inclusion lactateH12 : arterial lactate level at 12h

SECONDARY OUTCOMES:
Tissue oxygenation 6 | 6 hours
  Percentage of patients with normal arterial lactate level at 6 hours (<=2 mmol/L) or a relative decrease (or clearance) of arterial lactate level above 30% according to the formula (lactateH0 - lactateH6)/lactate H0*100.
  lactateH0 : arterial lactate level at inclusion lactateH6 : arterial lactate level at 6h
Tissue oxygenation 24 | 24 hours
  Percentage of patients with normal arterial lactate level at 24 hours (<=2 mmol/L) or a relative decrease (or clearance) of arterial lactate level above 30% according to the formula (lactateH0 - lactateH24)/lactate H0*100.
  lactateH0 : arterial lactate level at inclusion lactateH24 : arterial lactate level at 24h
Tissue oxygenation 48 | 48 hours
  Percentage of patients with normal arterial lactate level at 48 hours (<=2 mmol/L) or a relative decrease (or clearance) of arterial lactate level above 30% according to the formula (lactateH0 - lactateH48)/lactate H0*100.
  lactateH0 : arterial lactate level at inclusion lactateH48 : arterial lactate level at 48h
Mortality 7 | 7 days
  Percentage of Death at 7 days
Mortality 28 | 28 days
  Percentage of Death at 28 days
ICU mortality | 28 days
  Percentage of Death in ICU at 28 days
Hospital mortality | 28 days
  Percentage of Death in Hospital at 28 days
Change in SOFA 24 | 24 hours
  Differences between SOFA score at inclusion (SOFA0) and SOFA score at 24 hours. The sequential organ failure assessment score (SOFA score) ranges from 0 (normal patient) to 24 (most severe patient).
  Vincent JL, de Mendonça A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998;26(11):1793-800.
Change in SOFA 48 | 48 hours
  Differences between SOFA score at inclusion (SOFA0) and SOFA score at 48 hours. The sequential organ failure assessment score (SOFA score) ranges from 0 (normal patient) to 24 (most severe patient).
  Vincent JL, de Mendonça A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998;26(11):1793-800.
Change in SOFA 72 | 72 hours
  Differences between SOFA score at inclusion (SOFA0) and SOFA score at 72 hours. The sequential organ failure assessment score (SOFA score) ranges from 0 (normal patient) to 24 (most severe patient).
  Vincent JL, de Mendonça A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998;26(11):1793-800.
Change in SOFA 7d | 7 days
  Differences between SOFA score at inclusion (SOFA0) and SOFA score at day 7. The sequential organ failure assessment score (SOFA score) ranges from 0 (normal patient) to 24 (most severe patient).
  Vincent JL, de Mendonça A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998;26(11):1793-800.
ventilator free days | 28 days
  ventilator free days (VFDs) are defined as follows: VFDs=0: If the patient dies before 28 days. VFDs=(28-x): If the patient is success-fully weaned from mechanical ventilation within 28 days, where x is the number of days spent receiving mechanical ventilation.
  VFDs=0: If the patient requires mechanical ventilation for 28 days or more.
vasopressor free days | 28 days
  vasopressor free days (VaFDs) are defined as follows: VaFDs=0: If the patient dies before 28 days. VaFDs=(28-x): If the patient is successfully weaned from vasopressor within 28 days, where x is the number of days spent with vasopressor.
  VaFDs=0: If the patient requires vasopressor for 28 days or more.
renal replacement therapy free days | 28 days
  renal replacement therapy free days (RRFDs) are defined as follows: RRFDs=0: If the patient dies before 28 days. RRFDs=(28-x): If the patient is successfully weaned from renal replacement therapy within 28 days, where x is the number of days spent with vasopressor.
  RRFDs=0: If the patient requires renal replacement therapy for 28 days or more.
ICU length of stay | 28 days
  time spent in ICU from inclusion censored at 28 days
Ischemic | 28 days
  Incidence of ischemic event during the first 28 days (stroke, myocardial infarction, mesenteric infarction)
thrombosis | 28 days
  Incidence of deep venous thrombosis or pulmonary embolism during the first 28 days
TRIALI | 28 days
  Incidence of transfusion-related acute lung injury during the first 28 days
Transfusion reaction | 28 days
  Incidence of side effects of transfusions during the first 28 days (fever, chills, hemolysis)

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Amiens Picardie Site Sud, Amiens
  - Hopital Robert Ballanger, Aulnay-sous-Bois
  - Hopital Avicenne AP-HP, Bobigny
  - CH sud-Francilien, Corbeil
  - Hopital Henri Mondor AP-HP, Créteil
  - CHV André Mignot, Le Chesnay
  - Salengro, CHRU, Lille
  - CH Lyon Sud, Lyon
  - GH Édouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - GH Sud Ile de France, Melun
  - Bel Air CHR, Metz
  - Mercy, CHR, Metz
  - CHU de Nantes, Nantes
  - La Source, CHR, Orléans
  - Hopital Cochin AP-HP, Paris
  - Hopital de La Pitié Salpetriere AP-HP, Paris
  - Hopital Saint Antoine AP-HP, Paris
  - Hopital Saint Louis AP-HP, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided